CLINICAL TRIAL: NCT01078766
Title: Constraint-induced Movement Therapy and Hand Arm Bimanual Training in Children With Hemiplegic CP
Brief Title: Constraint-induced Movement Therapy and Hand Arm Bimanual Training in Children With Hemiplegic Cerebral Palsy (CP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 920090440
Record Dates: First submitted 2010-02-28; First posted 2010-03-02 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2015-06

CONDITIONS: Cerebral Palsy; Hand Function
Keywords: cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CIMT+HABIT (Experimental): Form of "summer camp", for six hours per day for 10 consecutive work days.
  Interventions: Other: CIMT+HABIT

INTERVENTIONS:
Other: CIMT+HABIT — The daily schedule included one hour of constraining the functional arm with intensive activation of the hemi-paretic arm and then 5 hours of various structured, intensive bimanual functional activities,

SUMMARY:
The combination of the constraint-induced movement therapy (CIMT) method as a complement to hand arm bimanual training (HABIT) will improve the frequency and quality of cooperative hand use and function in children with hemiplegic CP.

ELIGIBILITY:
Inclusion Criteria:

* active wrist extension/dorsiflexion of at least 20;
* MACS 1-3;
* GMFCS 1-2;
* enrolled in regular or remedial level education with ability to understand instructions and participate without parent presence.

Exclusion criteria:

* seizures;
* severely increased muscle tone; or hemi arm to good;
* orthopedic surgery on the upper extremity;
* botulin toxin injections within the past half year to the upper extremity;
* inability to understand instructions or cognitive/behavior/concentration.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment | twice before the intervention: one month and two days before as control period, and three times after the intervention: within the last two days, two months and six months after the end of the intervention program
  Rasch built, it measures how effectively a child with unilateral disability typically makes use of their affected (assisting) hand during bimanual performance. It is conducted by a semi-structured play session requiring bimanual handling that is video-recorded. Scoring is performed by a analyzing the video on 22 predefined items using a 4-point criterion-referenced rating scale

SECONDARY OUTCOMES:
Jebsen-Taylor Test of Hand Function | twice before the intervention: one month and two days before as control period, and three times after the intervention: within the last two days, two months and six months after the end of the intervention program
The Pediatric Evaluation of Disability Inventory (PEDI) | twice before the intervention: one month and two days before as control period, and three times after the intervention: within the last two days, two months and six months after the end of the intervention program
Muscle strength | twice before the intervention: one month and two days before as control period, and three times after the intervention: within the last two days, two months and six months after the end of the intervention program